CLINICAL TRIAL: NCT04646499
Title: Feasibility of Gamma Transcranial Alternating Current Stimulation to Reduce Beta-amyloid Load and Improve Memory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 131887a; R21AG060335 (NIH)
Record Dates: First submitted 2020-11-10; First posted 2020-11-30 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Gamma Stimulation Group (Experimental): This group will receive gamma stimulation
  Interventions: Device: Transcranial alternating current stimulation

INTERVENTIONS:
Device: Transcranial alternating current stimulation — Transcranial alternating current stimulation (tACS) will be applied at 40 Hz (gamma band) during eight sessions over the course of a month.

SUMMARY:
This project assessed the feasibility of transcranial alternating current stimulation in the gamma band to lower beta-amyloid load and improve memory performance.

DETAILED DESCRIPTION:
Thirteen individuals with aMCI received eight 60-minute sessions of 40-Hz (gamma) transcranial alternating current stimulation (tACS) in a single-arm design. Outcome measures were assessed pre- and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Grade 12 or more education
* Normal or corrected to normal vision and hearing
* Ability to complete cognitive tasks
* Ability to cooperate and comply with all study procedures
* Ability to tolerate tACS
* Self-reported memory complaint
* Diagnosed with mild cognitive impairment
* Amyloid positive

Exclusion Criteria:

* Neurological or psychiatric disorders other than mild cognitive impairment
* Receiving investigational medications or have participated in a trial with investigational medications within last 30 days
* Family history of epilepsy
* Implanted electronic devices (e.g., pacemaker)
* Prior head trauma
* Pregnant
* IQ < 80
* Taking cholinesterase inhibitory, memantine, or psychotropic medication
* Taking anti-depressants or anti-anxiety medication
* Color blind
* Substance abuse
* Glaucoma
* Macular degeneration
* Amblyopia (lazy eye)
* Strabismus (crossed eyes)

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Zanto, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The dataset includes self-reported information, behavioral and electrophysiological data. The final dataset will be stripped of identifiers prior to release for sharing, thereby anonymizing the data. We will make the anonymized data available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to attempt to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. This will be in accordance with human subject regulations.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available after the results have been determined and the study researchers are unblinded. The data will be available indefinitely upon request.
Access Criteria: Contact PI.

RESULTS

PARTICIPANT FLOW:
Groups:
- Gamma Stimulation Group: This group received gamma stimulation
  Transcranial alternating current stimulation: Transcranial alternating current stimulation (tACS) was applied at 40 Hz (gamma band) during eight sessions over the course of a month.
Period: Overall Study
Arm/Group | Gamma Stimulation Group
Started | 14
Completed | 13
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gamma Stimulation Group
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] — One participant was enrolled, but dropped out prior to data collection. Population: Only data from participants who completed the full protocol were analyzed.
  years | 74 (5)
Sex: Female, Male [Count of Participants; unit: Participants] — One participant was enrolled, but dropped out prior to data collection. Population: Only data from participants who completed the full protocol were analyzed.
  Participants
    Female | 6
    Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: One participant was enrolled, but dropped out prior to data collection.
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 13
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One participant was enrolled, but dropped out prior to data collection.
  Participants
    American Indian or Alaska Native | 0
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 1
    White | 11
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: One participant was enrolled, but dropped out prior to data collection.
  Participants
    United States | 13
Beta Amyloid [Mean (Standard Deviation); unit: unitless ratio] — Plasma-based beta amyloid 42/40 ratio. Population: One participant was enrolled, but dropped out prior to data collection. Only data from participants who completed the full protocol were analyzed. Higher values indicate worse outcomes.
  unitless ratio | 0.06 (0.02)
Tau [Mean (Standard Deviation); unit: pg/mL] — Plasma-based measure of pTau181 Population: One participant was enrolled, but dropped out prior to data collection. Only data from participants who completed the full protocol were analyzed. Higher values indicate worse outcomes.
  pg/mL | 3.38 (0.97)
Memory: Recall [Mean (Standard Deviation); unit: number of items correctly remembered] — Short Delay Free Recall portion of the California Verbal Learning Test Population: One participant was enrolled, but dropped out prior to data collection. Only data from participants who completed the full protocol were analyzed.
  number of items correctly remembered | 6.54 (4.29)
Memory: Paired Associates [Mean (Standard Deviation); unit: percentage of items correctly remembered] — Population: One participant was enrolled, but dropped out prior to data collection. Only data from participants who completed the full protocol were analyzed.
  percentage of items correctly remembered | 60 (20)
Memory: Fluency [Mean (Standard Deviation); unit: number of items named] — Memory fluency was assessed via the FAS test. Population: One participant was enrolled, but dropped out prior to data collection. Only data from participants who completed the full protocol were analyzed. Higher is better. Unit is number of items named that start with the letter f, a, or s.
  number of items named | 14.67 (3.78)

OUTCOME MEASURES:

1. Primary Outcome: Side Effects
Description: Side effects were measured on a scale from 0 (not noticable) to 10 (not tolerable): headache, neck pain, scalp pain, tingling, itching, burning sensation, increased sleepiness, trouble concentrating, acute mood change, and phosphenes. Average rating across all measures reported as indicator of side effects.
Time Frame: Average of all post-tACS sessions, up to 1 month
Population: Only data from participants who completed the full protocol were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gamma Stimulation Group
Number analyzed (Participants) | 13
units on a scale | 0.53 (0.65)

2. Primary Outcome: Drop Out
Description: Drop out rate will be assessed as the number of participants who withdraw or are withdrawn from the study.
Time Frame: post-tACS, up to 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Gamma Stimulation Group
Number analyzed (Participants) | 14
Participants | 1

3. Secondary Outcome: Beta Amyloid Load Change
Description: Change in plasma-based beta amyloid (AB) load was assessed as the AB42/40 ratio, calculated as post minus pre AB42/40 ratio. Greater increase is better.
Time Frame: pre-tACS (baseline) and post-tACS (1 month)
Population: Only data from participants who completed the full protocol were analyzed.
Measure: Mean (Standard Deviation); unit: unitless ratio
Arm/Group | Gamma Stimulation Group
Number analyzed (Participants) | 13
unitless ratio | 0.0008 (0.006)
Statistical Analysis 1: Comparison: Gamma Stimulation Group; Test type: Superiority; p = 0.34, Sign test

4. Secondary Outcome: Memory: Recall Change
Description: Episodic memory was assessed pre and post intervention as the number of words correct during the short delay free recall portion of the California Verbal Learning Test. Change was assessed as post minus pre. Greater increase is better.
Time Frame: pre-tACS (baseline), post-tACS (after one month of treatment)
Population: Only data from participants who completed the full protocol were analyzed.
Measure: Mean (Standard Deviation); unit: words correct
Arm/Group | Gamma Stimulation Group
Number analyzed (Participants) | 13
words correct | 1.5 (2.1)
Statistical Analysis 1: Comparison: Gamma Stimulation Group; Test type: Superiority; p = 0.024, Sign test

5. Secondary Outcome: Memory: Paired Associates Change
Description: Episodic memory was assessed pre and post intervention from memory accuracy for a paired associates task for visual objects. Change was assessed post minus pre. Greater increase is better.
Time Frame: pre-tACS (baseline), post-tACS (after one month of treatment)
Population: Only data from participants who completed the full protocol were analyzed.
Measure: Mean (Standard Deviation); unit: percent correct
Arm/Group | Gamma Stimulation Group
Number analyzed (Participants) | 13
percent correct | 11.5 (21.0)
Statistical Analysis 1: Comparison: Gamma Stimulation Group; Test type: Superiority; p = 0.083, Sign test

6. Secondary Outcome: Memory: Fluency Change
Description: Episodic memory fluency was assessed pre and post intervention from performance on the FAS task. Unit of measurement is the number of words names starting with the letter f, a, or s. Change was calculated as post minus pre. Greater increase is better.
Time Frame: pre-tACS (baseline), post-tACS (after one month of treatment)
Population: Only data from participants who completed the full protocol were analyzed.
Measure: Mean (Standard Deviation); unit: number of items named
Arm/Group | Gamma Stimulation Group
Number analyzed (Participants) | 13
number of items named | 1.5 (2.6)
Statistical Analysis 1: Comparison: Gamma Stimulation Group; Test type: Superiority; p = 0.049, Sign test

7. Secondary Outcome: Change in Tau
Description: Plasma tau levels was assessed pre and post intervention. Change was calculated as post minus pre. Greater decrease is better.
Time Frame: pre-tACS (baseline), post-tACS (after one month of treatment)
Population: Only data from participants who completed the full protocol were analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Gamma Stimulation Group
Number analyzed (Participants) | 13
pg/mL | 0.27 (0.72)
Statistical Analysis 1: Comparison: Gamma Stimulation Group; Test type: Superiority; p = 0.31, Sign test

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Gamma Stimulation Group
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/99/NCT04646499/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/99/NCT04646499/ICF_001.pdf